CLINICAL TRIAL: NCT06502496
Title: Behavioural Study in Chronic Pain : Creativity and Motivation, and Circuits Involved in Functional MRI
Acronym: AART
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HBD_2023_8
Record Dates: First submitted 2024-07-09; First posted 2024-07-16 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Art Therapy

STUDY DESIGN:
Masking Description: In order to limit biases linked to the absence of blinding and to potential patient preferences for one or other of the interventions, a "consent to postponed information" type of consent (Boter et al. 2003) will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- art-therapy (Experimental): Art therapy workshops : groups of 6 to 12 patients supervised over a session of 1.5 to 2 hours, in the presence of an artist and the nursing staff (psychologist, nurse, doctor). There are 6 sessions per group, with an average of one week between sessions.
  Interventions: Behavioral: art-therapy
- relaxation (Active Comparator): Relaxation workshops (control group): groups of 6 to 12 patients supervised over a session of 1.5 to 2 hours, in the presence of the psychologist. 5 sessions per group, with an average of one week between sessions.
  Interventions: Behavioral: relaxation

INTERVENTIONS:
Behavioral: art-therapy — Over the 6 sessions, different artistic techniques will be explored, depending on the artist leading the workshop: stencil, graffiti, spray paint, collage, oil pastel, calligraphy and acrylic doodling. A collective work may also be proposed.
  Arms: art-therapy
Behavioral: relaxation — relaxation sessions with the referent psychologist
  Arms: relaxation

SUMMARY:
Being creative means having the ability to produce ideas, actions or works that are original and different from what we have already done. This process involves mental flexibility, in particular the association of distant ideas or divergent thinking. This creative potential is complex and depends on a number of factors, both internal (personality, motivation, emotional state, stress) and external to the individual (socio-cultural context). The generation of creative ideas involves the fronto-striatal circuit, with a balance between flexibility and perseverance. The striatum is central to the reward system and mental flexibility, while the prefrontal cortex is involved in executive control, underpinning perseverance functions. Dopamine plays a key role in this balance, and changes in dopamine levels, depending on the type of receptor activated, will have a direct impact on the transition between mental flexibility and perseverance. Furthermore, in the context of chronic pain, changes in connectivity and activity can be observed in neuroimaging in these same regions of the reward circuit. This suggests that the dopaminergic system is also involved in the chronicisation of pain. The creative process would therefore be correlated with the dopaminergic reward system, involving several dimensions, both cognitive in terms of mental flexibility, coping strategies and perseverance, and motivational. In this context, art therapy treatments are beginning to be studied, particularly in patients suffering from Alzheimer's or Parkinson's disease, showing improvements in anxiety and depression.

Art therapy has not yet been widely proposed or studied for patients suffering from chronic pain. A more detailed behavioural study would confirm and clarify the clinical benefits for patients, by exploring the neuronal circuits involved, particularly the dopaminergic reward system.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 and over
* Consent to participate in the study
* Available for protocol visits
* Treated for chronic pain

Exclusion Criteria:

* Progressive neurodegenerative neurological pathology impairing cognitive function
* Untreated clinical depressive syndrome
* Fibromyalgia in the foreground
* High doses of opioid treatment (greater than 100 mg/d of morphine equivalent)
* Impaired judgement or inability to receive information that prevents performance of behavioural tasks
* Absolute contraindication to MRI (e.g. pacemaker and implantable stimulator not MRI compatible, intra-orbital metallic foreign body);
* Persons benefiting from a legal protection measure
* Pregnant or breast-feeding women
* Patient deprived of liberty
* Patient suffering from mental disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
changes in performance to obtain a reward (reward-based learning task) between before the sessions and 1 to 2 weeks after the sessions | Day0 and 1 to 2 weeks after the last session
  the reward learning ability will be assessed using a specific task. The result of the task questionnaire is a numeric score.

IPD SHARING:
Plan to Share IPD: No